CLINICAL TRIAL: NCT06390306
Title: The Efficacy and Safety of Third Generation Tyrosine Kinase Inhibitors Combined With Azacitidine and B-cell Lymphoma-2 Inhibitor in Patients With Myeloid Blast Phase Chronic Myeloid Leukemia
Brief Title: The Efficacy and Safety of Third-generation TKIs Combined With Azacitidine and Bcl-2 Inhibitor in Patients With CML-MBP
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Henan Cancer Hospital (Other Government); Zhejiang University (Other); Peking Union Medical College (Other); Nanfang Hospital, Southern Medical University (Other); Beijing Chuiyangliu Hospital (Other Government)
Responsible Party: Principal Investigator, Qian Jiang, Professor, Peking University People's Hospital
Other Study IDs: 2023PHB323-002
Record Dates: First submitted 2024-04-18; First posted 2024-04-30 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — ponatinib; Azacitidine; venetoclax; olverembatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — blood, bone marrow
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 3G-TKI + AZA + Ven group: Adult CML-MBP
  Interventions: Drug: Ponatinib; Drug: Azacitidine; Drug: Venetoclax; Drug: Olverembatinib

INTERVENTIONS:
Drug: Ponatinib — Ponatinib is recommended orally (PO) daily continuously on days 1-28 in 28-day cycle. Treatment repeats every 28 days in the absence of disease progression, unacceptable toxicity or HSCT.
Drug: Azacitidine — Azacitidine is recommended 75mg/m2 subcutaneously on days 1-7 in 28-day cycle. Treatment repeats every 28 days in the absence of disease progression, unacceptable toxicity or HSCT.
Drug: Venetoclax — Venetoclax is recommended orally (PO) daily on days 1-14 in 28-day cycle. Treatment repeats every 28 days in the absence of disease progression, unacceptable toxicity or HSCT.
Drug: Olverembatinib — Olverembatinib is recommended orally (PO) every other day on days 1-28 in 28-day cycle. Treatment repeats every 28 days in the absence of disease progression, unacceptable toxicity or HSCT.

SUMMARY:
This is a prospective multi-center study to investigate efficacy and safety of the third generation tyrosine kinase inhibitors (TKIs) combined with azacitidine and B-cell lymphoma-2 (Bcl-2) inhibitor in patients with myeloid blast phase chronic myeloid leukemia (CML-MBP).

DETAILED DESCRIPTION:
CML-MBP has dismal outcome. Currently, there is no standardized induction treatment approach in CML-MBP. The European LeukemiaNet (ELN) recommendations and NCCN guideline recommended the combination of TKI and chemotherapy in CML-MBP. The previous study revealed that TKI combined with hypomethylating agents had promising efficacy. However, imatinib and second generation TKI are the most widely applied in combination treatment, there is limited data in third generation TKI.

Currently, venetoclax in combination with hypomethylating agents such as azacitidine is standard treatment for patients with AML unsuitable for intensive induction chemotherapy. Maiti et al. reported that TKI combined with venetoclax and detectable had promising efficacy in CML-MBP. Therefore, the investigator conducted a study to explore the efficacy and safety of a third generation TKI in combination with azacitidine and Bcl-2 inhibitor in CML-MBP and multi-omics exploratory analysis was performed to identify potential biomarkers correlated with the outcome.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years old;
2. philadelphia chromosome (Ph)-positive or BCR::ABL-positive;
3. serum creatinine ≤ 1.5 × upper limit of normal (ULN) or 24h creatinine clearance ≥ 50 mL/min when serum creatinine was > 1.5 × ULN;
4. serum total bilirubin ≤ 1.5 × ULN;
5. aspartate aminotransferase and alanine aminotransferase ≤ 2.5 × ULN;
6. amylase ≤ 1.5 × ULN; (7) lipase ≤ 1.5 × ULN;
7. ejection fraction > 50%; corrected QT interval on electrocardiographic evaluation was ≤ 450 ms in men or ≤ 470 ms in women.

Exclusion Criteria:

1. concurrent diseases requiring treatment(s) with potential to interact with 3G-TKI;
2. diagnosis of other primary malignancies;
3. history of allogeneic HSCT;
4. extramedullary disease only.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Peking universuty people's hospital Union Hospital, Tongji Medical College, Huazhong University of Science and Technology Henan Cancer Hospital The First Affiliated Hospital, Zhejiang University School of Medicine Chinese Academy of Medical Sciences & Peking Union Medical College Hospital Nanfang Hospital, Southern Medical University Chuiyangliu hospital affiliated to tsinghua university The First Affiliated Hospital of Nanjing Medical University Qilu Hospital of Shandong University Xi'an International Medical Center Hospital Nanyang Central Hospital Ningbo Medical Center Lihuili Hospital Beijing Lu Daopei Hospital Sichuan Provincial People's Hospital The First Affiliated Hospital of Kunming Medical University The First Affiliated Hospital of Guangxi Medical University
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Major hematologic response (MaHR) | At the end of Cycle 2 (each cycle is 28 days)
  either a complete hematologic response (CHR) or no evidence of leukemia (NEL).

SECONDARY OUTCOMES:
Return to chronic phase | At the end of Cycle 2 (each cycle is 28 days)
  < 10% blasts in blood and bone marrow with no extra-medullary leukemia and last for ≥ 4 weeks
Major cytogenetic response (MCyR) | Up to 3 years
  Ph-positive cells ≤ 35%
Complete cytogenetic response (CCyR) | Up to 3 years
  no Ph-positive cell
Major molecular response (MMR) | Up to 3 years
  BCR::ABL1IS ≤ 0.1%
Event-free survival (EFS) | Up to 3 years
  interval from therapy start to lacking RCP after 1 cycle, MaHR after 2 cycles, loss of hematologic response, progression to blast phase again, or death from any causes
CML-related survival | Up to 3 years
  interval from therapy start to death from blast phase, or censored at the last follow-up
Survival | Up to 3 years
  interval from therapy start to death from any cause or censored at the last follow-up
Incidence of adverse events | Up to 3 years
  Adverse effects (AEs) were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0. and assessed continuously.

CONTACTS AND LOCATIONS:
Overall Officials: Qian Jiang, MD, Principal Investigator — Peking University People's Hospital
Locations (15):
- China (15):
  - Peking university people's hospital, Beijing, Beijing Municipality
  - Beijing Lu Daopei Hospital, Beijing
  - Chuiyangliu hospital affiliated to tsinghua university, Beijing
  - Sichuan Provincial People's Hospital, Chengdu
  - Nanfang Hospital, Southern Medical University, Guangdong
  - The First Affiliated Hospital of Kunming Medical University, Kunming
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Nanyang Central Hospital, Nanyang
  - Ningbo Medical Center Lihuili Hospital, Ningbo
  - Qilu Hospital of Shandong University, Qilu
  - Chinese Academy of Medical Sciences & Peking Union Medical College Hospital, Tianjin
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology Henan Cancer Hospital, Wuhan
  - Xi'an International Medical Center Hospital, Xi'an
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Zhejiang

IPD SHARING:
Plan to Share IPD: No